CLINICAL TRIAL: NCT01446380
Title: Phenotypic Expressions in a French Pseudoxanthoma-Elasticum Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC 2008 871
Record Dates: First submitted 2010-02-03; First posted 2011-10-05 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Pseudoxanthoma Elasticum
MeSH Terms: conditions — Pseudoxanthoma Elasticum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sera,Plasma,DNA,skin biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pseudoxanthoma elasticum

SUMMARY:
The cohort is intended to study the phenotypic expressions of the pseudoxanthoma elasticum (PXE) disease in various tissues (eye, skin, arteries, etc).

DETAILED DESCRIPTION:
This national french cohort is intended to improve our knowledge on the PXE disease. The study of phenotypic expression of the diseases is focused on cutaneous, opthalmologic and vascular tissues. All investigations are included in a yearly follow-up for these patients and collected in a database.

Plasma are also collected for all patients and stored in our clinical research biological center in Angers, including genetic (DNA) material extracted from diagnostic skin biopsy. French Ministry of Teaching and Research Authorisation number for the PXE collection is AC 2008 871. Declarative number is DC 2008 870.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PXE disease
* Informed consent obtained
* Patient affiliated to Health care system (french social security)

Exclusion Criteria:

* No informed consent
* No affiliation to a Health care system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed for a PXE disease from any part of France and requesting a follow-up and clinical management of there disease (opthalmic and vascular complications mainly).
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2008-06; Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic MARTIN, MD PhD, Study Director — UH Angers
Locations (1):
- University Hospital of Angers, Angers, Pays de Loire, France

REFERENCES:
- [Background] Naouri M, Boisseau C, Bonicel P, Daudon P, Bonneau D, Chassaing N, Martin L. Manifestations of pseudoxanthoma elasticum in childhood. Br J Dermatol. 2009 Sep;161(3):635-9. doi: 10.1111/j.1365-2133.2009.09298.x. Epub 2009 Jun 9. PMID 19519828
- [Background] Martin L, Maitre F, Bonicel P, Daudon P, Verny C, Bonneau D, Le Saux O, Chassaing N. Heterozygosity for a single mutation in the ABCC6 gene may closely mimic PXE: consequences of this phenotype overlap for the definition of PXE. Arch Dermatol. 2008 Mar;144(3):301-6. doi: 10.1001/archderm.144.3.301. PMID 18347285
- [Derived] Biere L, Donal E, Terrien G, Furber A, Martin L, Prunier F. Left ventricular function in a large cohort of pseudoxanthoma elasticum patients. PLoS One. 2014 Mar 20;9(3):e90364. doi: 10.1371/journal.pone.0090364. eCollection 2014. PMID 24651258